CLINICAL TRIAL: NCT03494465
Title: Randomised Controlled Trial to Evaluate the Efficacy and Safety of Lens Extraction in Patients With Pseudoexfoliation Glaucoma: a Feasibility and Pilot Study
Brief Title: Efficacy and Safety of Lens Extraction in Patients With Pseudoexfoliation Glaucoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xerencia de Xestión Integrada de Ferrol (Other)
Responsible Party: Principal Investigator, SARA POSE BAZARRA, Ophthalmologist, MD, Xerencia de Xestión Integrada de Ferrol
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FACOPEX
Record Dates: First submitted 2018-03-21; First posted 2018-04-11 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Pseudoexfoliation Glaucoma; Intraocular Pressure
MeSH Terms: conditions — Exfoliation Syndrome | interventions — Phacoemulsification

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MEDICAL TREATMENT GROUP (Active Comparator): Medical treatment will be used in a staggered manner and may also associate laser trabeculoplasty. If necessary, then surgical treatment would be indicated: trabeculectomy. or another filtering surgery.
  Inadequate IOP control will be determined by the local ophthalmologist, and additional treatment will be indicated to achieve an target IOP.
  Interventions: Drug: MEDICAL GLAUCOMA TREATMENT
- INTERVENTION GROUP (Experimental): In lens extraction arm, patients will undergo lens phacoemulsification with intraocular lens implant (IOL) within 60 days after randomization.
  If additional treatment is required, the same stepped sequence of therapy described for "medical treatment group" will be used and will be considered a therapeutic failure.
  Interventions: Procedure: PHACOEMULSIFICATION

INTERVENTIONS:
Procedure: PHACOEMULSIFICATION — Standard phacoemulsification with intraocular lens implant will be perform within 60 days after allocation. If IOP target is not achieve, patients will be treated as in "medical treatment group"
  Arms: INTERVENTION GROUP
Drug: MEDICAL GLAUCOMA TREATMENT — The escalation of topical hypotensive medications will be carried out with the following sequence: 1. single topical medication; 2. double topical therapy; 3. triple topical therapy. Beginning, with the exception of individual contraindications, with prostaglandin analogs, followed by topical beta-blockers, carbonic anhydrase inhibitors and finally alpha-agonists.Target IOP will be used in both groups to inform the need of escalation of therapy; in patients with ocular hypertension the target IOP will be 21 mmHg. In patients with mild glaucoma target IOP will be 18 mmHg, and in patients with moderate glaucoma the target IOP will be 15 mmHg.
  Arms: MEDICAL TREATMENT GROUP

SUMMARY:
There are several publications that have demonstrated the protective role of cataract surgery against the development of long-term glaucoma, especially in cases of pseudoexfoliation glaucoma (PXFG). Cataract surgery in patients with pseudoexfoliation (PXF) is a procedure with higher rates of complications due to its smaller pupillary diameter and its greater zonular weakness, so lens extraction performed earlier could possibly reduce intra and postoperative complications. Given the severity and high prevalence of PXFG in our environment, investigators proposed a randomized clinical trial to evaluate the efficacy of cataract surgery in reducing the intraocular pressure (IOP) at 12 months and thereby change the course of the disease. The control group will have glaucoma treatment according to standard practice.

DETAILED DESCRIPTION:
INTRODUCTION

Pseudoexfoliation (PXF) is a pathology characterized by the accumulation of extracellular microfibrillar material in the anterior segment of the eye. It was first described by Lindberg in Finland in 1917 and is the most common identifiable cause of glaucoma. It is diagnosed clinically with the observation of a white-greyish fibrillar material mainly on the anterior surface of the lens, but also in the pupillary margin or other ocular tissues, as well as in other structures: blood vessels, skin, kidneys, heart, lungs or meninges, among others. It is considered a multifactorial disease that involves genetic and non-genetic factors and whose pathogenesis is based on the theory of microfibrillar elastosis, creating an excessive amount of pseudoexfoliative material that aggregates, deposits and increases resistance in the trabecular meshwork, with the consequent increase of intraocular pressure (IOP).

According to the World Health Organization, glaucoma is the leading cause of irreversible blindness in the world. Pseudoexfoliative glaucoma (PXFG) is the second most frequent subtype of glaucoma, after primary open-angle glaucoma (POAG). Its incidence increases progressively with age and the prevalence varies between countries, being estimated in the area under investigation around 6.5%, increasing to 28.3% in patients over 80 years. Its prognosis is more severe than in POAG, and the risk of developing glaucoma is between 5 and 10 times more frequent in eyes with PXF.

The current medical management for PXFG is similar to POAG, beginning with medical therapy. Sometimes it can also be associated with laser treatment, trabeculoplasty, which is effective only in the short term. As the last step we resort to glaucoma surgery, trabeculectomy, or other filtering surgeries, which have a variable success rate, and although the efficacy is similar to those of POAG, complications are more frequent in this type of patients.

There are multiple publications that have demonstrated the protective role of cataract surgery in the long-term development of glaucoma, especially in PXFG cases. It was also described a moderate reduction in IOP after phacoemulsification in PXF patients, but noted that there is still insufficient scientific evidence for more severe glaucoma or poor IOP control. This reduction in intraocular pressure seems to be maintained over time, even 7 years after the extraction of the cataract.

In addition, there is evidence that eyes with PXF benefit especially from cataract surgery and reduce the risk of glaucoma. Although cataract surgery in patients with PXF is a procedure with higher complication rates due to its smaller pupillary diameter and its greater zonular weakness, a lens surgery performed earlier (non-hypermature cataracts or scarce dilatations) could reduce possible intra- and post-operative complications. It has been reported that the highest incidence of complications appears in patients who show signs of zonular weakness, so this type of patients will not be included in this study in order to avoid possible relative complications. On the other hand, an increase in the incidence of complications has been reported in relation to later ages at the time of cataract surgery, therefore earlier surgery would imply a possible decrease in long-term complications with an improvement in the quality of life of patients.

Regarding the studies mentioned on cataract and PXF surgery, investigators did not find references on the BCVA preoperative. The indication for cataract surgery is based on the presence of a surgical cataract without determining any visual acuity limit. The patients that are proposed to be included in the study are patients who present cataracts, with ages over 60 years and pseudoexfoliation and suffering from glaucoma or ocular hypertension. Investigators will limit the best-corrected visual acuity (BCVA) to less than 0.7 (decimal scale) as long as there are visual symptoms due to the presence of the cataract, such as photophobia, difficulties in activities of daily living or driving, but with BVCA greater than or equal to 0.4 in order not to recruit mature cataracts and thereby reduce possible intra- and post-operative complications.

In the experience in routine practice clinicians have seen patients with PXFG who have benefited from lens extraction while maintaining well-controlled IOP values over time. It is also part of the usual clinic to indicate surgery in patients with PXFG in which a mild-moderate IOP reduction can be achieve with a safer surgery than trabeculectomy. There is no randomized study or protocol that indicates when surgery is most effective or when it would be more beneficial for both, the patient and the health care system. Taking into account that they are patients who usually undergo this type of surgery, it seems necessary to carry out a randomized clinical study that allows us to objectify our hypothesis.

Due to the severity of PXFG and its high prevalence in the environment under investigation, researchers propose this pilot study to evaluate the hypothesis that PXFG could be treated earlier with lens surgery and thereby change the course of the disease. Cataract surgery is an effective and safe procedure with great potential, since it is a simple intervention that can substantially improve the quality of life of patients and improve the control of intraocular pressure.

TARGET POPULATION

The study will be carried out with patients recruited from the public health care system (SERGAS) in the Ophthalmology Units of the Hospital University Complex of Ferrol and Santiago de Compostela

RANDOMIZATION

Patients will be randomized in two groups in equal proportion (1:1 ratio) by using opaque envelopes due to the small sample size to obtain the same proportion in both treatment groups.

A. Medical Treatment Group B. Intervention group

SAMPLE SIZE

Calculation of the sample size is carried out to estimate the minimum number of participants needed to detect a significant statistical result, and it depends in part on the value of the standard deviation (SD). This SD is usually unknown. Clinical trials with few patients can provide imprecise estimates. In general, investigators should take into account the ability to evaluate and include patients and also consider the likelihood of specifying the effects of treatment.

According to the papers published by Sim & Lewis and Hertzog, sample sizes between 24 and 50 participants have been recommended for clinical feasibility studies. Consequently, researchers consider that a sample of between 40 and 50 patients can give a precise and concrete vision of the aims the investigators intend to achieve. It is based on the calculation of the confidence interval as 1.96 x √ (p x (1-p) / n), where p is the percentage that is expected to be seen, and n is the size of the sample. Investigators will therefore relate the sample size with a confidence interval of 95%.

One of the aims of this RCT is to be able to estimate an SD that allow to calculate the sample size of a long-term multicentre randomized clinical trial, in addition to the participation, abandonment and compliance rate.

MEASUREMENTS AND INTERVENTIONS

Two ophthalmologists (SPB and MJVL), one per centre, will perform the lens extraction surgeries. A standardized surgical protocol will be agreed between both surgeons. The calculation of the biometric power will be made with an IOL Master (Carl Zeiss Meditec), and the formula SRK-T will be used. For eyes with less than 22 mm axial length, another additional formula, the Hoffer Q, will be used for comparative purposes. The refraction aim will depend on the eye.

IOP measurement (primary outcome) will be masked by using a second observer to perform the IOP measurement.

Goldman or Perkins applanation tonometer will be used to check IOP.

Humphrey Perimeter (Threshold test strategy: SITA Standard 24-2) (Carl Zeiss Meditec) will be used for monitoring visual fields.

The reliability of the visual field will be determined by: percentage of false negatives <15%, percentage of false positives <15% and percentage of loss of fixation <15%. The global indexes are numerical parameters that summarize the results of the visual fields. The most useful index is the MD (mean deviation) that represents the average difference between the normal sensitivity corrected by age, and the measurement of the threshold values at each point of the test.

RNFL determinations will be carried out with the OCT Heidelberg (Heidelberg Engineering Spectralis®) and the "Glaucoma Module Premium Edition" program provides an analysis of the nerve fiber layer of the retina (RNFL) through an anatomical scan of the optic nerve head.

The best-corrected visual acuity will be taken on the Snellen scale with the optotypes adjusted to the patient's focal distance.

Pachymetry: It will be taken by ultrasonic pachymetry equipment, the gold standard.

Biomicroscopy and funduscopy will be visualized by slit lamp.

Quality of visual function: a quality of life questionnaire will be carried out, VFQ-25 Visual Functioning Questionnaire 25 (NIE VFQ 25 National Eye Institute Visual Function Quality 25) before randomization and once the study is completed in order to objectify the improvements in the visual quality of patients after lens extraction.

Cataract surgery is an outpatient procedure that does not require admission or hospital stays, as well as glaucoma filtering surgeries. Participants who undergo cataract extraction will sign a informed consent which is the same used in daily clinical practice, detailing the specific risks of PXF syndrome, in the same way that it has been carried out as an usual practice.

Economic analysis. Cost-benefit analysis: this trial aims to evaluate the feasibility of a definitive randomized controlled trial (RCT) comparing PXFG medical treatment versus cataract extraction. The economic aspect serves as a tool to determine the most efficient therapeutic method at public health care system, taking into account the use of resources that include the costs of the interventions and the pharmacological cost. It is expected that the main cost factor of the cataract surgery group is itself and the components include staff, anesthesia, consumables in surgery and the costs of the intervention will be obtained from the costs of SERGAS. The cost derived from medical treatment will be originated mainly from eye drops. The costs of these drugs are public knowledge. Costs derived from other types of interventions, mainly glaucoma filtering surgery, will also be obtained from the budgets provided by SERGAS

INTERVENTION DESCRIPTION

Visit 1: Information. Proposal to participate in the study and signing the informed consent. Randomization

Visit 2: Complete examination (BCVA, IOP, biomicroscopy, funduscopy, OCT NRFL). Pachymetry and first visual field test to be included in the pretreatment study. Questionnaire VFQ25. IOL master biometry.

Visit 2: Intervention arm: Cataract surgery will be performed within 60 days of randomization. Postoperative visits will be done at first day, first week and at first month.

Control visits: 3 visits will be schedule every 4 months until complete 12 months (complete examination will be performed) According to the individual requirements and at the ophthalmologist's decision, more visits may be made for better control and management of glaucoma.

Last visit: Complete exploration, VFQ25 questionnaire and final visual field test.

STATISTICAL ANALYSIS

Statistical analysis as well as the graphical results will be carried out with professional statistical software (SPSS). A descriptive analysis of the clinical variables will be carried out. The continuous variables will be expressed as mean and standard deviation and the categorical variables as number of cases and percentages.

A single main statistical analysis will be carried out at the end of the trial when every follow-up has been completed. The results listed above will be compared between both groups (intervention group and control group) using linear models (analysis of covariance). The statistical significance will be adjusted to the level of 5% (p <0.05).

The quality of life will be evaluated with visual function quality questionnaires (VFQ25) and the unit of analysis will be the participant / patient. The analysis of subgroups in terms of the main outcome (IOP) will be carried out according to the randomization group (intervention group / control group).

SAFETY

The possible complications related to cataract surgery will be the same as in standardized cataract surgeries for all other patients:

* Expulsive hemorrhage
* Endophthalmitis
* Opacity of the anterior and posterior capsule
* Damage of the posterior capsule
* Pseudophakic macular edema
* Retinal detachment
* Dislocation/luxation of the intraocular lens

In addition, eyes with PXF present a higher risk of complications during cataract surgery such as zonular detachment, posterior capsule rupture or insufficient pupillary dilation, but also greater long-term risks such as opacification of the posterior capsule or subluxation of the lens complex. However, lens extraction in patients with early PXF may be safer and technically less difficult than in patients with more advanced PXF and cataracts, since less ultrasonic power is required for phacoemulsification, less manipulation during surgery, and less postoperative inflammation.

One of the most frequent late postoperative complications is the dislocation of the IOL complex, and as described in the meta-analysis of Vázquez-Ferreiro et al there is no greater incidence of subluxations with time after surgery (average range 5.5-8.5 years), although it has been related to elderly patients at the time of cataract surgery or previous zonular weakness. Therefore, early surgery would mean a possible reduction in long-term complications.

This type of patients is currently undergoing cataract surgery with the same indications as in cases in which there is no PXF as part of the clinical practice. The study aims to minimize the possible complications related to surgery, recruiting patients with a higher safety profile, excluding those patients who show signs of zonular weakness, pupil dilation less than 5mm or hypermature/mature cataracts.

ETHICAL-LEGAL ASPECTS

The development of the project will be carried out respecting the Declaration of Helsinki of the World Medical Association 1964 and successive ratifications on ethical principles for medical research in human beings; and the Oviedo Convention for the protection of human rights and the dignity of the human being with respect to the applications of Biology and Medicine, made on April 4, 1997, ratified by Spain on July 23, 1999 and successive updates.

The researchers are familiar with the protocol and with the data collection. The essential documents will be maintained to demonstrate the validity of the study and the integrity of the collected data. The master files will be constituted at the beginning of the study, will be maintained during their realization and will be conserved according to the applicable regulations. The Research Ethics Committee (CEI) will review all relevant study documentation in order to safeguard the rights, safety and well being of patients. The study will only be carried out at the centre where the CEI authorization has been obtained.

The researchers participating in this study agree that any clinical data collected from the subjects to be studied should be separated from the personal identification data, guaranteeing the confidentiality of the participants in the research and respecting the Law of Protection of Personal Data (Organic Law 15/1999, of December 13) and Royal Decree 1720/2007, of December 21, which approves the Development Regulation of this law, Law 41/2002, of November 14 (basic regulatory of the patient's autonomy and of rights and obligations in terms of information and clinical documentation), as well as Law 3/2001, of May 28 (regulating the informed consent and the clinical history of patients), Law 3/2005, of March 7, modification of Law 3/2001 and Decree 29/2009 of February 5, which regulates access to electronic medical records.

The researchers will collect the clinical data of the patients to the study in the Data Collection Notebook (DCN). Each DCN will be coded, protecting the patient's identity. Only the research team and the health authorities, which have a duty to maintain confidentiality, will have access to all the data collected for the study and will keep the file that relates codes with identification data. Only information that can not be identified will be transmitted to third parties (the code file will not be sent, only the non-identifiable data will be sent). Once the study is finished, the data will be anonymized for future use, requesting express permission for this in the informed consent for the participants.

ECONOMIC SUMMARY

No financial support is required for the execution of this project, so the economic memory of this project is 0 euros. This study has not been funded, and neither patients nor researchers charge for participation in it.

ELIGIBILITY:
Inclusion criteria:

1. Presence of cataract with visual symptoms that justify the intervention, such as photophobia, difficulty in activities of daily living or driving.
2. Mild or moderate PXF glaucoma or ocular hypertension (OHT) over 25mmHg + PXF syndrome.

   Glaucoma is defined as: reproducible defects (two or more contiguous points with a loss of P <0.01, three or more contiguous points with a loss of P <0.05 or greater) in the visual field (VF) or , ophthalmoscopically detectable damage to the optic nerve (cup disc ratio> or = 0.7 and / or focal thinning of the optic nerve rim and / or asymmetry of cup disc ratio > or = 0.2 between both eyes).

   PXF is defined clinically by the presence of pseudoexfoliative material in the anterior capsule of the lens.

   Mild glaucoma is defined as MD< 6dB. Moderate glaucoma is defined as MD < 12dB.
3. Naive patients or without topical hypotensive treatment in the last 3 months.
4. Age: patients > 60 years.
5. Best corrected visual acuity (BCVA) between range > 0.4 and <0.7
6. Signature of the specific informed consent of the study.

Exclusion criteria:

1. Advanced glaucoma. It is defined as an average deviation > -15dB and / or threat of fixation (paracentral point with sensitivity of 0 dB), and / or cup disc ratio > 0.9
2. Corneal edema, corneal opacity or any other known corneal factor that may increase the risk of complications during surgery
3. Previous cataract surgery in the eye included in the study
4. Axial length <20 mm
5. Estimated IOL power> 30 diopters
6. Visual acuity <0.4 or> 0.7
7. Signs of zonular weakness: phacodonesis, iridodonesis, lens subluxation, asymmetry of anterior chamber depth
8. Pupillary dilation <5 mm
9. Advanced cataract

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2021-03-28 (Actual)

PRIMARY OUTCOMES:
INTRAOCULAR PRESSURE | 12 months
  The primary outcome will be the intraocular pressure (IOP) reduction 12 months after randomisation

SECONDARY OUTCOMES:
VISUAL FIELD INDEX | 12 months
  Visual field (VF) progression according to the global VF index (VFI) at 12 months
RETINAL NERVE FIBER LAYER | 12 months
  Retinal nerve fiber layer (RNFL) thickness by optical coherence tomography (OCT): investigators will compare the reduction in the retinal nerve fiber layer by OCT according to the premium analysis of glaucoma (Heidelberg) between both arms of the treatment at 12 months
INCIDENCE OF GLAUCOMA SURGERY | 12 months
  Number of trabeculectomy or filtering surgery required as a result of poor control of IOP or progression in the VF in both groups at 12 months
BEST CORRECTED VISUAL ACUITY | 12 months
  Best-corrected visual acuity (BCVA): investigators will compare the change of visual acuities (VA) between randomisation and last follow-up at 12 months.
QUALITY OF LIFE. VFI Q25 CUESTIONAIRE | 12 months
  Investigators will evaluate changes in quality of life before and 12 months after the intervention, using a visual function quality questionnaire: National Eye Institute Visual Function Questionnaire (NEI-VFQ25).
  Translation of the 2000 version of the National Eye Institute Visual Function Quality -25, public domain will be used. (Mangione CM, Lee PP, Gutierrez PR, Spritzer K, Berry S, Hays RD, National Eye Institute Visual Function Questionnaire Field Test Investigators, Development of the 25-item National Eye Institute Visual Function Questionnaire, Arch Ophthalmol, 2001 Jul; 119 ( 7): 1050-8.)
NUMBER OF GLAUCOMA DRUGS | 12 months
  Number of glaucoma drugs as well as the possible intolerances to it: Investigate the reduction of drugs after cataract surgery and the adverse effects of these in patients who require topical treatment. Comparison of both groups in search of better quality of life and tolerance of both treatments.
COST BENEFIT ANALYSIS | 12 months
  Through a cost-benefit analysis investigators will evaluate the common and pertinent costs in each treatment arm and evaluate the health benefit in economic terms
INCIDENCE OF TREATMENT ADVERSE EVENTS | 12 months
  Investigators will determine the safety profile of both interventions through an evaluation of intraoperative and post-treatment complications
RATE OF RECRUITMENT | 12 months
  To estimate rates of recruitment among eligible patients who are offered trial participation, and withdrawal rates to confirm the feasibility of conducting a large and definite randomized clinical trial to evaluate cataract surgery as a treatment for patients with PXFG.

CONTACTS AND LOCATIONS:
Locations (1):
- Sara Pose-Bazarra, Ferrol, A Coruna, Spain

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Ritch R. Exfoliation syndrome. Curr Opin Ophthalmol. 2001 Apr;12(2):124-30. doi: 10.1097/00055735-200104000-00008. PMID 11224719
- [Background] Schlotzer-Schrehardt U, Naumann GO. Ocular and systemic pseudoexfoliation syndrome. Am J Ophthalmol. 2006 May;141(5):921-937. doi: 10.1016/j.ajo.2006.01.047. PMID 16678509
- [Background] Streeten BW, Gibson SA, Dark AJ. Pseudoexfoliative material contains an elastic microfibrillar-associated glycoprotein. Trans Am Ophthalmol Soc. 1986;84:304-20. PMID 3590474
- [Background] Viso E, Rodriguez-Ares MT, Gude F. Prevalence of pseudoexfoliation syndrome among adult Spanish in the Salnes eye Study. Ophthalmic Epidemiol. 2010 Mar;17(2):118-24. doi: 10.3109/09286581003624970. PMID 20302433
- [Background] Kristianslund O, Ostern AE, Raen M, Sandvik GF, Drolsum L. Does cataract surgery reduce the long-term risk of glaucoma in eyes with pseudoexfoliation syndrome? Acta Ophthalmol. 2016 May;94(3):261-5. doi: 10.1111/aos.12945. Epub 2016 Jan 9. PMID 26749122
- [Background] Chen PP, Lin SC, Junk AK, Radhakrishnan S, Singh K, Chen TC. The Effect of Phacoemulsification on Intraocular Pressure in Glaucoma Patients: A Report by the American Academy of Ophthalmology. Ophthalmology. 2015 Jul;122(7):1294-307. doi: 10.1016/j.ophtha.2015.03.021. Epub 2015 May 2. PMID 25943711
- [Background] Moghimi S, Johari M, Mahmoudi A, Chen R, Mazloumi M, He M, Lin SC. Predictors of intraocular pressure change after phacoemulsification in patients with pseudoexfoliation syndrome. Br J Ophthalmol. 2017 Mar;101(3):283-289. doi: 10.1136/bjophthalmol-2016-308601. Epub 2016 Jun 8. PMID 27281754
- [Background] Vazquez-Ferreiro P, Carrera-Hueso FJ, Poquet Jornet JE, Fikri-Benbrahim N, Diaz-Rey M, Sanjuan-Cervero R. Intraoperative complications of phacoemulsification in pseudoexfoliation: Metaanalysis. J Cataract Refract Surg. 2016 Nov;42(11):1666-1675. doi: 10.1016/j.jcrs.2016.09.010. PMID 27956295
- [Background] Shingleton BJ, Neo YN, Cvintal V, Shaikh AM, Liberman P, O'Donoghue MW. Outcome of phacoemulsification and intraocular lens implantion in eyes with pseudoexfoliation and weak zonules. Acta Ophthalmol. 2017 Mar;95(2):182-187. doi: 10.1111/aos.13110. Epub 2016 May 27. PMID 27230126
- [Background] Astrom S, Stenlund H, Linden C. Intraocular pressure changes over 21 years - a longitudinal age-cohort study in northern Sweden. Acta Ophthalmol. 2014 Aug;92(5):417-20. doi: 10.1111/aos.12232. Epub 2013 Jul 31. PMID 23902137
- [Background] Mitchell P, Wang JJ, Hourihan F. The relationship between glaucoma and pseudoexfoliation: the Blue Mountains Eye Study. Arch Ophthalmol. 1999 Oct;117(10):1319-24. doi: 10.1001/archopht.117.10.1319. PMID 10532440
- [Background] Chang RT, Shingleton BJ, Singh K. Timely cataract surgery for improved glaucoma management. J Cataract Refract Surg. 2012 Oct;38(10):1709-10. doi: 10.1016/j.jcrs.2012.08.030. No abstract available. PMID 22999597
- [Background] Pohjalainen T, Vesti E, Uusitalo RJ, Laatikainen L. Intraocular pressure after phacoemulsification and intraocular lens implantation in nonglaucomatous eyes with and without exfoliation. J Cataract Refract Surg. 2001 Mar;27(3):426-31. doi: 10.1016/s0886-3350(00)00691-x. PMID 11255056
- [Background] Ekstrom C, Botling Taube A. Pseudoexfoliation and cataract surgery: a population-based 30-year follow-up study. Acta Ophthalmol. 2015 Dec;93(8):774-7. doi: 10.1111/aos.12789. Epub 2015 Jun 11. PMID 26095907
- [Background] Mamalis N. Exfoliation syndrome: effects of cataract surgery on glaucoma. J Cataract Refract Surg. 2008 Nov;34(11):1813-4. doi: 10.1016/j.jcrs.2008.09.002. No abstract available. PMID 19006713
- [Background] Vazquez-Ferreiro P, Carrera-Hueso FJ, Fikri-Benbrahim N, Barreiro-Rodriguez L, Diaz-Rey M, Ramon Barrios MA. Intraocular lens dislocation in pseudoexfoliation: a systematic review and meta-analysis. Acta Ophthalmol. 2017 May;95(3):e164-e169. doi: 10.1111/aos.13234. Epub 2016 Aug 29. PMID 27569700
- [Background] Jakobsson G, Zetterberg M, Lundstrom M, Stenevi U, Grenmark R, Sundelin K. Late dislocation of in-the-bag and out-of-the bag intraocular lenses: ocular and surgical characteristics and time to lens repositioning. J Cataract Refract Surg. 2010 Oct;36(10):1637-44. doi: 10.1016/j.jcrs.2010.04.042. PMID 20870107
- [Background] Shingleton BJ, Laul A, Nagao K, Wolff B, O'Donoghue M, Eagan E, Flattem N, Desai-Bartoli S. Effect of phacoemulsification on intraocular pressure in eyes with pseudoexfoliation: single-surgeon series. J Cataract Refract Surg. 2008 Nov;34(11):1834-41. doi: 10.1016/j.jcrs.2008.07.025. PMID 19006727
- [Background] Zetterstrom C, Behndig A, Kugelberg M, Montan P, Lundstrom M. Changes in intraocular pressure after cataract surgery: analysis of the Swedish National Cataract Register Data. J Cataract Refract Surg. 2015 Aug;41(8):1725-9. doi: 10.1016/j.jcrs.2014.12.054. PMID 26432131
- [Background] Poley BJ, Lindstrom RL, Samuelson TW, Schulze R Jr. Intraocular pressure reduction after phacoemulsification with intraocular lens implantation in glaucomatous and nonglaucomatous eyes: evaluation of a causal relationship between the natural lens and open-angle glaucoma. J Cataract Refract Surg. 2009 Nov;35(11):1946-55. doi: 10.1016/j.jcrs.2009.05.061. PMID 19878828
- [Background] Elgin U, Sen E, Simsek T, Tekin K, Yilmazbas P. Early Postoperative Effects of Cataract Surgery on Anterior Segment Parameters in Primary Open-Angle Glaucoma and Pseudoexfoliation Glaucoma. Turk J Ophthalmol. 2016 Jun;46(3):95-98. doi: 10.4274/tjo.92604. Epub 2016 Jun 6. PMID 27800269
- [Background] Sim J, Lewis M. The size of a pilot study for a clinical trial should be calculated in relation to considerations of precision and efficiency. J Clin Epidemiol. 2012 Mar;65(3):301-8. doi: 10.1016/j.jclinepi.2011.07.011. Epub 2011 Dec 9. PMID 22169081
- [Background] Hertzog MA. Considerations in determining sample size for pilot studies. Res Nurs Health. 2008 Apr;31(2):180-91. doi: 10.1002/nur.20247. PMID 18183564